CLINICAL TRIAL: NCT00165789
Title: A Randomized, Double Blind, Placebo Controlled, Parallel Group Study to Explore the Safety And Tolerability of Doses of E2007 Up to a Maximum of 8 mg In Patients With Parkinson's Disease Who Experience End-of-Dose Wearing Off Motor Fluctuations
Brief Title: A Study to Explore the Safety And Tolerability of Doses of E2007 Up to a Maximum of 8 mg In Patients With Parkinson's Disease Who Experience End-of-Dose Wearing Off Motor Fluctuations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: E2007-A001-214
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Results first posted 2015-06-02 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-04

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — perampanel

INTERVENTIONS:
Drug: E2007

SUMMARY:
This is a randomized, double-blind, two treatment, two group, parallel group study. Subjects will be randomized to one of two treatment groups (E2007 or Placebo) in a 3 to 1 ratio and receive treatment for a total of ten weeks (Days 1 to 70).

ELIGIBILITY:
Inclusion Criteria:

* Subjects of any race greater than or equal to 30 years of age
* Have a diagnosis of idiopathic Parkinson's disease. Subjects should fulfill the UK Parkinson's Disease Society Brain Bank Clinical Diagnostic criteria (Queen Square criteria) and have a rating of 2 - 4 on the Hoehn and Yahr scale when in an 'off' state.
* Receiving an optimized regimen of anti-Parkinsonian treatments that has been stable for at least four weeks before baseline. The regimen is not considered to be stable if "as required" or "on demand" dosing is routinely used or there is regular use of apomorphine or liquid forms of levodopa.
* Taking levodopa or levodopa-containing medications (e.g. co-beneldopa, cocareldopa) at least three times daily with a good response to each levodopa dose as evidenced from patient diaries or medical notes.
* Consistently experience end-of-dose "wearing-off" motor fluctuations. Subjects should:
* score greater than or equal to 1 on Question 39 (What proportion of the waking day is the patient "off" on average?) of the full UPDRS at screening.
* have at least 2.5 hours of "off" time on average per day recorded in the patient diary at baseline.
* Willing and able to provide written informed consent and adhere to the protocol requirements, including completion of a patient diary.

Exclusion Criteria:

* Receiving treatment with medication known to induce CYP3A4 activity
* Previous stereotactic surgery (e.g. pallidotomy, subthalamic nucleus deep brain stimulation) for Parkinson's disease
* Received an investigational product within four weeks prior to screening or having participated in a previous study with E2007.
* Clinically significant cognitive impairment [mini-mental state examination (MMSE) less than 24 or fulfilling DSM IV criteria for dementia due to Parkinson's disease].
* Active hepatic disease, significantly reduced hepatic function or significantly elevated liver enzymes (abnormal bilirubin or serum transaminase levels of more than 1.5 times the upper limit of the normal range).
* Clinically significant ECG abnormality, including prolonged QTc (defined as QTc greater than or equal to 450 msec for males and greater than or equal to 470 msec for females using Fridericia's correction).
* Clinically significant, cardiovascular, metabolic, respiratory, renal, endocrinological, gastrointestinal diseases, psychiatric disorders, and bacterial or viral infections within the previous 30 days.
* History of drug or alcohol abuse.
* Women who are pregnant or lactating.
* Any condition that could, in the opinion of the investigator, place the subject at increased risk or is likely to prevent completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2005-09; Primary Completion 2006-02 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Arroyo, M.D., Ph.D, Study Director — Eisai Inc.
Locations (10):
- United States (10):
  - Clinical Trials Incorporated, Little Rock, Arkansas
  - UMDNJ - Robert Wood Johnson Medical School, Oxnard, California
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, New Haven, Connecticut
  - Inc., Boca Raton, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Suncoast Neuroscience Associates, St. Petersburg, Florida
  - Raleigh Neurology Associates, Southfield, Michigan
  - Agape Medical Research Center, Piscataway, New Jersey
  - Inc., Raleigh, North Carolina
  - The Clinical Neuroscience Center, Lubbock, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 - Placebo; Cohort 2- Placebo: Placebo matching Perampanel dosing once daily for 10 weeks.
- Cohort 1 - Perampanel: Perampanel started at 2 mg once daily for 2 weeks, followed by 3 mg once daily for 2 weeks, followed by 4 mg once daily for 2 weeks, followed by 6 mg once daily for 4 weeks.
- Cohort 2 - Perampanel: Perampanel started at 2 mg once daily for 2 weeks, followed by 4 mg once daily for 2 weeks, followed by 6 mg once daily for 2 weeks, followed by 8 mg once daily for 4 weeks.
Period: Overall Study
Arm/Group | Cohort 1 - Placebo | Cohort 1 - Perampanel | Cohort 2- Placebo | Cohort 2 - Perampanel
Started | 8 | 20 | 12 | 35
Completed | 8 | 16 | 11 | 21
Not Completed | 0 | 4 | 1 | 14
Not completed — Adverse Event | 0 | 3 | 0 | 12
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Cohort 2 - Placebo: Placebo matching Perampanel dosing once daily for 10 weeks.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - Placebo | Cohort 1 - Perampanel | Cohort 2 - Placebo | Cohort 2 - Perampanel | Total
Number analyzed (Participants) | 8 | 20 | 12 | 35 | 75
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.6 (10.43) | 68.5 (7.78) | 68.5 (12.71) | 67.5 (10.48) | 68.025 (10.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 10 | 3 | 11 | 26
  Male | 6 | 10 | 9 | 24 | 49

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline to Day 70 in "on" State of UPDRS Scores
Description: The Unified Parkinson's Disease Rating Scale (UPDRS) consisted of 4 subsections used to assess symptoms and signs of Parkinson's disease, with an overall scale range of 0-147. Individual subsections included: I. Mentation, behavior, and mood (0-16); II. Activities of daily living assessed in both the "on" and "off" state (0-52); III. Motor examination (0-56); and IV. Complications of therapy assessed in the "on" fluctuations and dyskinesias (0-23). Each subsection included subscales that ranged from 0 (best possible outcome) to 1 or 4 (worst possible outcome), with the total score of subsection equaling the sum of the scores of the subscales and the overall UPDRS score equaling the sum of the scores of the 4 subsections (higher score indicating more severe Parkinson's Disease).
Time Frame: Baseline and Day 70
Population: Safety Population. Change from Baseline only reflect participants who completed the assessment at Baseline and Day 70.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Cohort 1 - Placebo | Cohort 1 - Perampanel | Cohort 2 - Placebo | Cohort 2 - Perampanel
Number analyzed (Participants) | 8 | 15 | 11 | 21
Scores on a Scale
  Overall Score | -7.13 (13.601) | -5.33 (6.355) | -1.18 (10.806) | 0.05 (7.117)
  Mentation, Behavior, and Mood | -0.88 (0.641) | 0 (1.134) | -0.73 (1.104) | 0.86 (1.526)
  Activities of Daily Living | 0.75 (5.751) | -0.27 (3.615) | 1 (4.648) | 0.24 (2.755)
  Motor Examinations | -6.38 (9.149) | -3.93 (5.365) | -0.73 (5.587) | -1.14 (5.452)
  Complications of Therapy | -0.63 (4.241) | -1.13 (1.685) | -0.73 (3.467) | 0.1 (2.663)

2. Secondary Outcome: Change From Baseline to Day 70 in Absolute "Off" Time
Description: Subjects and/or caregiver completed a diary recording their motor state and dyskinesia symptoms over the course of the day before and at the end of study drug dosing on 3 consecutive days leading up to Baseline and Day 70. An entry was made every 30 minutes whether they were in the "on" state experiencing troubling dyskinesias or "off" state. The "on" state reflected recovery of control of a particular Parkinsonian feature that readily responded to each dose of levodopa, while the "off" state reflected the re-emergence of that feature. Troublesome dyskinesias were unintentional movements that occurred while in the "on" state and which interfered with activities or caused discomfort to any extent.
Time Frame: Baseline and Day 70
Population: Safety Population. Change from Baseline only reflect participants who completed the assessment at Baseline and Day 70.
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Cohort 1 - Placebo | Cohort 1 - Perampanel | Cohort 2 - Placebo | Cohort 2 - Perampanel
Number analyzed (Participants) | 8 | 15 | 11 | 20
Hour | -0.94 (2.162) | -2.11 (3.714) | -1.27 (2.411) | -0.93 (2.28)

3. Secondary Outcome: Change From Baseline to Day 70 in Absolute "on" Time With Non-troublesome Dyskinesias
Description: as for outcome 2
Time Frame: Baseline and Day 70
Population: Safety Population. Change from Baseline only reflect participants who completed the assessment at Baseline and Day 70.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Cohort 1 - Placebo | Cohort 1 - Perampanel | Cohort 2 - Placebo | Cohort 2 - Perampanel
Number analyzed (Participants) | 8 | 15 | 11 | 20
Hours | 0 (2.372) | -0.51 (1.634) | -0.14 (1.38) | 0.4 (1.536)

4. Secondary Outcome: Change From Baseline to Day 70 in Absolute "on" Time With Troublesome Dyskinesias
Description: as for outcome 2
Time Frame: Baseline and Day 70
Population: Safety Population. Change from Baseline only reflect participants who completed the assessment at Baseline and Day 70.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Cohort 1 - Placebo | Cohort 1 - Perampanel | Cohort 2 - Placebo | Cohort 2 - Perampanel
Number analyzed (Participants) | 8 | 15 | 11 | 20
Hours | -0.96 (1.471) | 0.57 (1.635) | -0.14 (1.074) | -0.48 (2.104)

5. Secondary Outcome: Change From Baseline to Day 70 in Goetz/Rush Score
Description: The Goetz/Rush scale was used to rate severity during performance of tasks intended to elicit dyskinesias, and provided an objective rating of dyskinesias during activities of daily living.The tasks included a sitting exercise, mental calculations, drinking, dressing, and walking. A 5-point scale was used: 0=absent; 1=minimal severity, no interference with voluntary motor acts; 2=dyskinesias, may impair voluntary movements but the subject was capable of efficiently completing the motor task; 3=intense dyskinesias, interference with movement control and completion of the motor task was greatly limited; 4= violent dyskinesias, incompatible with the completion of the motor task. A lower score indicated less difficulty performing the tasks.
Time Frame: Baseline and Day 70
Population: Safety Population. Change from Baseline only reflect participants who completed the assessment at Baseline and Day 70.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Cohort 1 - Placebo | Cohort 1 - Perampanel | Cohort 2 - Placebo | Cohort 2 - Perampanel
Number analyzed (Participants) | 8 | 16 | 11 | 21
Scores on a Scale | -1.63 (2.875) | 0.63 (1.784) | -0.3 (1.79) | -0.4 (1.77)

6. Secondary Outcome: Change From Baseline to Day 70 in Percent "Off" Time
Description: as for outcome 2
Time Frame: Baseline and Day 70
Population: Safety Population. Change from Baseline only reflect participants who completed the assessment at Baseline and Day 70.
Measure: Mean (Standard Deviation); unit: Percentage of the Day
Arm/Group | Cohort 1 - Placebo | Cohort 1 - Perampanel | Cohort 2 - Placebo | Cohort 2 - Perampanel
Number analyzed (Participants) | 8 | 15 | 11 | 20
Percentage of the Day | -7.46 (14.614) | -13.91 (23.06) | -7.9 (15.114) | -6 (12.388)

7. Secondary Outcome: Change From Baseline to Day 70 in Percent "on" Time
Description: as for outcome 2
Time Frame: Baseline and Day 70
Population: Safety Population. Change from Baseline only reflect participants who completed the assessment at Baseline and Day 70.
Measure: Mean (Standard Deviation); unit: Percentage of the Day
Arm/Group | Cohort 1 - Placebo | Cohort 1 - Perampanel | Cohort 2 - Placebo | Cohort 2 - Perampanel
Number analyzed (Participants) | 8 | 15 | 11 | 20
Percentage of the Day | -6.77 (10.408) | 3.07 (9.006) | -0.74 (5.792) | -3.16 (12.953)

8. Secondary Outcome: Change From Baseline to Day 70 in Percent "on" Time With Non-troublesome Dyskinesias
Description: as for outcome 2
Time Frame: Baseline and Day 70
Population: Safety Population. Change from Baseline only reflect participants who completed the assessment at Baseline and Day 70.
Measure: Mean (Standard Deviation); unit: Percentage of the Day
Arm/Group | Cohort 1 - Placebo | Cohort 1 - Perampanel | Cohort 2 - Placebo | Cohort 2 - Perampanel
Number analyzed (Participants) | 8 | 15 | 11 | 20
Percentage of the Day | 0.28 (15.672) | -2.49 (9.603) | -0.63 (7.653) | 2.75 (9.935)

9. Secondary Outcome: Disability of Dyskinesia From UPDRS at Baseline and Day 70
Description: The disability of dyskinesia was determined from question 33 (part 4) of the UPDRS assessment. It asks how disabling are the dyskinesias, and uses a 5-part scale: 0=Not disabling, 1=MIldly disabling, 2=Moderately disabling, 3=Severely disabling, 4=Completely disabling. Lower scores represented more normal functioning.
Time Frame: Baseline and Day 70
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Cohort 1 - Placebo | Cohort 1 - Perampanel | Cohort 2 - Placebo | Cohort 2 - Perampanel
Number analyzed (Participants) | 8 | 20 | 12 | 35
Participants
  Baseline, Not Disabling (n=8,20,12,35) | 5 | 13 | 8 | 18
  Baseline, Mildly Disabling (n=8,20,12,35) | 1 | 3 | 1 | 13
  Baseline, Moderately Disabling (n=8,20,12,35) | 1 | 2 | 3 | 2
  Baseline, Severely Disabling (n=8,20,12,35) | 0 | 2 | 0 | 1
  Baseline, Completely Disabling (n=8,20,12,35) | 1 | 0 | 0 | 0
  Day 70, Not Disabling (n=8,16,11,21) | 6 | 10 | 6 | 14
  Day 70, Mildly Disabling (n=8,16,11,21) | 1 | 3 | 4 | 3
  Day 70, Moderately Disabling (n=8,16,11,21) | 0 | 2 | 1 | 4
  Day 70, Severely Disabling (n=8,16,11,21) | 1 | 1 | 0 | 0
  Day 70, Completely Disabling (n=8,16,11,21) | 0 | 0 | 0 | 0

10. Secondary Outcome: Duration of Dyskinesia From UPDRS at Baseline and Day 70
Description: The duration of dyskinesia was determined from question 32 (part 4) of the UPDRS assessment. It asks what proportion of the waking day are dyskinesias present, and uses a 5-part scale: 0 = None, 1 = 1-25% of day, 2 = 26-50% of day, 3 = 51-75% of day, 4 = 76-100% of day. Lower scores represented more normal functioning.
Time Frame: Baseline and Day 70
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Cohort 1 - Placebo | Cohort 1 - Perampanel | Cohort 2 - Placebo | Cohort 2 - Perampanel
Number analyzed (Participants) | 8 | 20 | 12 | 35
Participants
  Baseline, None (n=8,20,12,35) | 1 | 5 | 4 | 11
  Baseline, 1 to 25% of Day (n=8,20,12,35) | 3 | 7 | 3 | 15
  Baseline, 26 to 50% of Day (n=8,20,12,35) | 3 | 3 | 4 | 6
  Baseline, 51 to 75% of Day (n=8,20,12,35) | 0 | 5 | 1 | 1
  Baseline, 76 to 100% of Day (n=8,20,12,35) | 1 | 0 | 0 | 1
  Day 70, None (n=8,16,11,21) | 1 | 6 | 4 | 7
  Day 70, 1 to 25% of Day (n=8,16,11,21) | 5 | 5 | 5 | 9
  Day 70, 26 to 50% of Day (n=8,16,11,21) | 2 | 4 | 2 | 5
  Day 70, 51 to 75% of Day (n=8,16,11,21) | 0 | 1 | 0 | 0
  Day 70, 76 to 100% of Day (n=8,16,11,21) | 0 | 0 | 0 | 0

11. Primary Outcome: Number of Participants With Any TEAE
Description: Treatment-emergent Adverse Events (TEAEs) were defined as those adverse events (AEs) that started on or after the first dose of study medication until the end of the study. Information on any AEs were recorded throughout the study after informed consent had been signed and included abnormal clinical laboratory tests, vital sign measurements and physical examinations. Note: Safety/tolerability info captured in Adverse Event section.
Time Frame: Through end of study
Population: Safety Population was the primary population for analysis defined as all subjects who completed the Baseline Phase and who received at least 1 dose of double-blind study medication.
Measure: Number; unit: Participants
Arm/Group | Cohort 1 - Placebo | Cohort 1 - Perampanel | Cohort 2 - Placebo | Cohort 2 - Perampanel
Number analyzed (Participants) | 8 | 20 | 12 | 35
Participants | 7 | 18 | 8 | 32

ADVERSE EVENTS:
Arm/Group | Cohort 1 - Placebo | Cohort 1 - Perampanel | Cohort 2 - Placebo | Cohort 2 - Perampanel
Serious Adverse Events (participants affected / at risk) | 0/8 | 4/20 | 0/12 | 4/35
Other Adverse Events (participants affected / at risk) | 7/8 | 18/20 | 8/12 | 32/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - Placebo (N=8) | Cohort 1 - Perampanel (N=20) | Cohort 2 - Placebo (N=12) | Cohort 2 - Perampanel (N=35)
FALL (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
ELECTROCARDIOGRAM ABNORMAL (Investigations) | 0 | 0 | 0 | 1
HEMIPARESIS (Nervous system disorders) | 0 | 0 | 0 | 1
PARKINSON'S DISEASE (Nervous system disorders) | 0 | 0 | 0 | 1
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 0 | 0 | 1
INSOMNIA (Psychiatric disorders) | 0 | 0 | 0 | 1
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - Placebo (N=8) | Cohort 1 - Perampanel (N=20) | Cohort 2 - Placebo (N=12) | Cohort 2 - Perampanel (N=35)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 1 | 0 | 0
ATRIAL FLUTTER (Cardiac disorders) | 1 | 0 | 0 | 0
ATRIOVENTRICULAR BLOCK FIRST DEGREE (Cardiac disorders) | 0 | 0 | 1 | 1
PALPITATIONS (Cardiac disorders) | 1 | 0 | 0 | 1
SUPRAVENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 0 | 1 | 0 | 0
TACHYCARDIA (Cardiac disorders) | 1 | 0 | 0 | 0
EAR DISCOMFORT (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
EAR PAIN (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
VERTIGO (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
LACRIMATION INCREASED (Eye disorders) | 0 | 1 | 0 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 | 0 | 0 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 1 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 0 | 1 | 0 | 1
DYSPHAGIA (Gastrointestinal disorders) | 0 | 1 | 0 | 0
GASTRITIS ATROPHIC (Gastrointestinal disorders) | 0 | 1 | 0 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 0 | 1 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 1 | 0 | 0
HIATUS HERNIA (Gastrointestinal disorders) | 0 | 1 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 4 | 0 | 2
VOMITING (Gastrointestinal disorders) | 0 | 2 | 0 | 2
ASTHENIA (General disorders) | 0 | 1 | 1 | 2
DIFFICULTY IN WALKING (General disorders) | 0 | 1 | 0 | 0
FATIGUE (General disorders) | 0 | 0 | 1 | 1
GAIT DISTURBANCE (General disorders) | 0 | 1 | 0 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 1 | 0 | 0 | 0
OEDEMA PERIPHERAL (General disorders) | 0 | 1 | 0 | 0
DENTAL CARIES (Infections and infestations) | 0 | 1 | 0 | 0
HELICOBACTER INFECTION (Infections and infestations) | 0 | 1 | 0 | 0
LARYNGITIS (Infections and infestations) | 1 | 0 | 0 | 0
NASOPHARYNGITIS (Infections and infestations) | 0 | 1 | 0 | 1
SINUSITIS (Infections and infestations) | 1 | 0 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 1 | 2 | 2 | 2
CONTUSION (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 2
FALL (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 3
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
BLOOD CHOLESTEROL INCREASED (Investigations) | 0 | 1 | 0 | 0
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 0 | 2 | 1 | 0
BLOOD CREATININE INCREASED (Investigations) | 0 | 1 | 0 | 0
BLOOD PRESSURE DECREASED (Investigations) | 0 | 0 | 1 | 2
BLOOD PRESSURE INCREASED (Investigations) | 0 | 0 | 1 | 1
ELECTROCARDIOGRAM CHANGE (Investigations) | 0 | 0 | 1 | 0
ELECTROCARDIOGRAM ST SEGMENT DEPRESSION (Investigations) | 0 | 1 | 0 | 0
HEART RATE INCREASED (Investigations) | 0 | 1 | 1 | 0
URINARY CASTS (Investigations) | 0 | 1 | 0 | 0
URINE LEUKOCYTE (Investigations) | 0 | 1 | 0 | 0
WHITE BLOOD CELLS URINE POSITIVE (Investigations) | 0 | 1 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2
MUSCLE RIGIDITY (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
POSTURE ABNORMAL (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
TENDONITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
BALANCE DISORDER (Nervous system disorders) | 1 | 2 | 0 | 1
BRADYKINESIA (Nervous system disorders) | 0 | 1 | 0 | 0
CHOREA (Nervous system disorders) | 0 | 1 | 0 | 0
DISTURBANCE IN ATTENTION (Nervous system disorders) | 0 | 1 | 0 | 0
DIZZINESS (Nervous system disorders) | 1 | 4 | 1 | 10
DIZZINESS POSTURAL (Nervous system disorders) | 0 | 0 | 2 | 0
DROOLING (Nervous system disorders) | 0 | 1 | 0 | 0
DYSGEUSIA (Nervous system disorders) | 0 | 1 | 0 | 0
DYSKINESIA (Nervous system disorders) | 1 | 2 | 0 | 2
DYSTONIA (Nervous system disorders) | 0 | 1 | 0 | 2
HEADACHE (Nervous system disorders) | 0 | 0 | 1 | 3
HYPERREFLEXIA (Nervous system disorders) | 0 | 1 | 0 | 0
MUSCLE SPASTICITY (Nervous system disorders) | 0 | 1 | 0 | 0
NYSTAGMUS (Nervous system disorders) | 0 | 0 | 1 | 1
PARKINSON'S DISEASE (Nervous system disorders) | 1 | 1 | 1 | 5
SEDATION (Nervous system disorders) | 0 | 0 | 0 | 4
SOMNOLENCE (Nervous system disorders) | 2 | 5 | 3 | 11
TREMOR (Nervous system disorders) | 1 | 1 | 1 | 0
TUNNEL VISION (Nervous system disorders) | 1 | 0 | 0 | 0
ABNORMAL DREAMS (Psychiatric disorders) | 1 | 0 | 0 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 1 | 0 | 2
DELUSION (Psychiatric disorders) | 0 | 2 | 0 | 0
DEPRESSION (Psychiatric disorders) | 0 | 1 | 1 | 0
HALLUCINATION,VISUAL (Psychiatric disorders) | 0 | 1 | 0 | 1
IMPULSIVE BEHAVIOUR (Psychiatric disorders) | 0 | 1 | 0 | 0
INITIAL INSOMNIA (Psychiatric disorders) | 0 | 0 | 1 | 0
INSOMNIA (Psychiatric disorders) | 0 | 2 | 1 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
SKIN LESION (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
SWELLING FACE (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
HYPERTENSION (Vascular disorders) | 0 | 0 | 0 | 2
HYPOTENSION (Vascular disorders) | 0 | 1 | 1 | 3
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1 | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No